CLINICAL TRIAL: NCT03256396
Title: Intraoperative Positive End-Expiratory Pressure Setting Guided By Esophageal Pressure Measurement in Patients Undergoing Laparoscopic Gynecologic Surgery
Brief Title: Intraoperative PEEP Setting During Laparoscopic Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Annop Piriyapatsom, MD, Lecturer, Department of Anesthesiology, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 253/2560(EC3)
Record Dates: First submitted 2017-08-11; First posted 2017-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Positive-Pressure Respiration/Methods; Esophagus/Physiopathology; Pleura/Physiopathology; Gynecologic Surgical Procedures; Laparoscopy; Humans; Female
Keywords: Intraoperative mechanical ventilation; Positive-end expiratory pressure; Esophageal pressure; Transpulmonary pressure; Laparoscopic gynecologic surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental): PEEP set according to esophageal pressure measured
  Interventions: Procedure: PEEP setting based on esophageal pressure measured
- Group C (No Intervention): PEEP set at 5 cm H2O

INTERVENTIONS:
Procedure: PEEP setting based on esophageal pressure measured — PEEP is set on the basis of esophageal pressure measurement with the aim to maintain transpulmonary pressure during expiration between 0 and 5 cmH2O
  Arms: Group E

SUMMARY:
The creation of pneumoperitoneum during laparoscopic surgery can have significant effects on the respiratory system including decreased respiratory system compliance, decreased vital capacity and functional residual capacity and atelectasis formation. Intraoperative mechanical ventilation, especially setting of positive end-expiratory pressure (PEEP) has an important role in respiratory management during laparoscopic surgery. The aim of this study is to determine whether setting of PEEP guided by measurement of pleural pressure would improve oxygenation and respiratory system compliance during laparoscopic surgery.

DETAILED DESCRIPTION:
As minimally invasive procedure with numerous advantages compared with open surgery, laparoscopic surgery has been substantially performed worldwide. The creation of pneumoperitoneum during laparoscopic surgery, however, can have significant effects on the respiratory system including decreased respiratory system compliance, decreased vital capacity and functional residual capacity and atelectasis formation. These pathophysiologic changes may put patients at risk of postoperative pulmonary complications. Therefore, intraoperative mechanical ventilation, especially setting of positive end-expiratory pressure (PEEP) has an important role in respiratory management during laparoscopic surgery. Nevertheless, there is no consensus on the optimal PEEP level and the best method to set PEEP during laparoscopic surgery. In patients with acute respiratory distress syndrome, PEEP set according to pleural pressure measured by using esophageal balloon catheter significantly has beneficial effects in terms of oxygenation, compliance and possible mortality. The aim of this study is to determine whether setting of PEEP guided by measurement of pleural pressure would improve oxygenation and respiratory system compliance during laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age of equal or more than 18 years old undergoing laparoscopic gynecologic surgery with anticipated surgical duration of more than 2 hours

Exclusion Criteria:

* Patients with ASA physical status of equal or more than 3
* Patients with significant cardiovascular or respiratory diseases
* Patients with significant pathological lesion in pharynx and esophagus that preclude placement of esophageal balloon catheter
* Patients with contraindications for PEEP titration such as increased intracranial pressure or unstable hemodynamic
* Patients with arrhythmias
* Patients who refuse to provide written informed consent
* Patients undergoing surgery with duration of less than 2 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Difference in PaO2 between Group E and Group C | At 15 minutes after initiation of pneumoperitoneum
Difference in PaO2 between Group E and Group C | At 60 minutes after initiation of pneumoperitoneum
Difference in PaO2 between Group E and Group C | At 30 minutes after arrival in recovery room

SECONDARY OUTCOMES:
Difference in compliance of respiratory system between Group E and Group C | At 15 minutes and 60 minutes after initiation of pneumoperitoneum, and 30 minutes after arrival in recovery room
Difference in alveolar dead space to tidal volume ratio between Group E and Group C | At 15 minutes and 60 minutes after initiation of pneumoperitoneum, and 30 minutes after arrival in recovery room
Difference in hemodynamics between Group E and Group C | At 15 minutes and 60 minutes after initiation of pneumoperitoneum
Proportion of thoracoabdominal transmission of intraabdominal pressure | At 15 minutes and 60 minutes after initiation of pneumoperitoneum
Adverse respiratory events | During 72 hours postoperatively or until discharge from hospital
  Adverse respiratory events define as requirement of oxygen supplement after discharge from the recovery room, episodes of desaturation (SpO2 of less than 90%), now-onset respiratory infection, new infiltration on chest radiograph, or respiratory failure.
Length of hospital stay | Up to 30 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Annop Piriyapatsom, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelosi P, Foti G, Cereda M, Vicardi P, Gattinoni L. Effects of carbon dioxide insufflation for laparoscopic cholecystectomy on the respiratory system. Anaesthesia. 1996 Aug;51(8):744-9. doi: 10.1111/j.1365-2044.1996.tb07888.x. PMID 8795317
- [Background] Rauh R, Hemmerling TM, Rist M, Jacobi KE. Influence of pneumoperitoneum and patient positioning on respiratory system compliance. J Clin Anesth. 2001 Aug;13(5):361-5. doi: 10.1016/s0952-8180(01)00286-0. PMID 11498317
- [Background] Gallart L, Canet J. Post-operative pulmonary complications: Understanding definitions and risk assessment. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):315-30. doi: 10.1016/j.bpa.2015.10.004. Epub 2015 Oct 22. PMID 26643097
- [Background] Valenza F, Chevallard G, Fossali T, Salice V, Pizzocri M, Gattinoni L. Management of mechanical ventilation during laparoscopic surgery. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):227-41. doi: 10.1016/j.bpa.2010.02.002. PMID 20608559
- [Background] Park SJ, Kim BG, Oh AH, Han SH, Han HS, Ryu JH. Effects of intraoperative protective lung ventilation on postoperative pulmonary complications in patients with laparoscopic surgery: prospective, randomized and controlled trial. Surg Endosc. 2016 Oct;30(10):4598-606. doi: 10.1007/s00464-016-4797-x. Epub 2016 Feb 19. PMID 26895920
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Result] Meininger D, Byhahn C, Mierdl S, Westphal K, Zwissler B. Positive end-expiratory pressure improves arterial oxygenation during prolonged pneumoperitoneum. Acta Anaesthesiol Scand. 2005 Jul;49(6):778-83. doi: 10.1111/j.1399-6576.2005.00713.x. PMID 15954959
- [Result] Maracaja-Neto LF, Vercosa N, Roncally AC, Giannella A, Bozza FA, Lessa MA. Beneficial effects of high positive end-expiratory pressure in lung respiratory mechanics during laparoscopic surgery. Acta Anaesthesiol Scand. 2009 Feb;53(2):210-7. doi: 10.1111/j.1399-6576.2008.01826.x. PMID 19175578
- [Result] Cinnella G, Grasso S, Spadaro S, Rauseo M, Mirabella L, Salatto P, De Capraris A, Nappi L, Greco P, Dambrosio M. Effects of recruitment maneuver and positive end-expiratory pressure on respiratory mechanics and transpulmonary pressure during laparoscopic surgery. Anesthesiology. 2013 Jan;118(1):114-22. doi: 10.1097/ALN.0b013e3182746a10. PMID 23196259
- [Result] Spadaro S, Karbing DS, Mauri T, Marangoni E, Mojoli F, Valpiani G, Carrieri C, Ragazzi R, Verri M, Rees SE, Volta CA. Effect of positive end-expiratory pressure on pulmonary shunt and dynamic compliance during abdominal surgery. Br J Anaesth. 2016 Jun;116(6):855-61. doi: 10.1093/bja/aew123. PMID 27199317
- [Derived] Piriyapatsom A, Phetkampang S. Effects of intra-operative positive end-expiratory pressure setting guided by oesophageal pressure measurement on oxygenation and respiratory mechanics during laparoscopic gynaecological surgery: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):1032-1039. doi: 10.1097/EJA.0000000000001204. PMID 32371830

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03256396/Prot_SAP_000.pdf